CLINICAL TRIAL: NCT05399173
Title: Effect of Laser Acupuncture for Treating Monosymptomatic Nocturnal Enuresis in Adolescent Females
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Jehan Hussien Mohammed Mustafa, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003689
Record Dates: First submitted 2022-05-23; First posted 2022-06-01 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Non-Specific Urethritis
Keywords: adolescents, nocturnal enuresis
MeSH Terms: conditions — Nocturnal Enuresis | interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- an infrared (gallium aluminum arsenide laser) (Experimental): Each female in study group will be treated by laser acupuncture for 3 sessions per week, for 6 weeks. An infrared (gallium aluminum arsenide) laser will be used at a wavelength of 808 nm and a power of 200 m W applied for 26 s to produce energy of less than 4 J/cm. participants will receive the same medical treatment (desmopressin acetate) and advice as in control group in addition to low level laser therapy 3 session / week for 6 weeks.
  Interventions: Device: infrared (gallium aluminum arsenide laser)
- conventional therapy (Active Comparator): They will receive medical treatment (desmopressin acetate) per-night dose of 120 g (for 6 weeks) & advice.
  Interventions: Drug: medical treatment(desmopressin acetate)

INTERVENTIONS:
Device: infrared (gallium aluminum arsenide laser) — Patient Position will be in supine & prone position, the area of these points is resolved utilizing anatomical landmarks and an arrangement of length measurements whose units are in respect to the physical extents of the individual patient. Acupuncture points used to treat nighttime enuresis are situated in regions that coincide with innervation by spinal sacral segments S2 through to S4 and expressed in the treatment conventions. The points of BL 23, BL 28, BL 32, RN 3, RN 4, RN 6, RN 12 impact the spinal micturition centers and parasympathetic innervation to the urinary tract, while excitement on scalp acupoints of DU 20 and DU 14 change cerebrum function through inner temporal, thalamencephalon and prefrontal cortical frameworks. Excitation of acupoints UB 20, UB 13, SP 6, ST 36, KI 3 and LU 9 are considered to strengthen spleen, vital energy and blood which encourage standardized bladder capacity
  Arms: an infrared (gallium aluminum arsenide laser)
Drug: medical treatment(desmopressin acetate) — participants will receive medical treatment (desmopressin acetate) per-night dose of 120 g (for 6 weeks) & advice
  Arms: conventional therapy

SUMMARY:
The aim of this study is to evaluate the effect of laser acupuncture on monosymptomatic nocturnal enuresis in adolescent females.

DETAILED DESCRIPTION:
Nocturnal enuresis (NE) can be defined as the involuntary passage of urine during sleep beyond the age of anticipated nighttime bladder control, which is generally accepted as 5 years of age.

IF neglected may persist into adulthood and be associated with urgency incontinence . It causes social, psychological, and emotional distress and carries a significant clinical burden. Studies show that enuretic children have lower self-esteem than healthy children. Even among chronic illnesses, enuresis has more negative effect on children's mental and social health .

Most of the studies highlighted that persisting NE was a high risk of psychosocial comorbidity and negatively affects the quality of life. The feeling of helplessness of enuretic patients highlights the magnitude and complexity of the problem. Persisting enuresis adversely affects the coping, social competence, and school performance of enuretic patients when compared to their normal peers. Furthermore, a negative correlation exists between the self-esteem of an enuretic child and the chance of treatment failure .

Complementary and alternative medicine (CAM) widely helped to encounter the increasing demand for non-pharmacological approaches. In recent years, there is a focus on finding cost-effective therapeutic approaches with minimal side effects to treat nocturnal enuresis .

Regarding the effect of laser acupuncture on nocturnal enuresis, previous studies about the effect of low level laser acupuncture on monosymptomatic nocturnal enuresis females are limited. There was only one previous study that examined the effect of low level laser acupuncture on bladder reservoir . This study will be the first one to objectively assess the effect of laser acupuncture in monosymptomatic nocturnal enuresis by sonography. As a result, this study will have variable benefits for medical care organizations and will add to the body of knowledge of physical therapists in the scientific domain. Control group will consist of 30 females. participants will receive medical treatment (desmopressin acetate, ) per-night dose of 120 g (for 6 weeks) & advice .

Study group will consist of 30 females. participants will receive the same medical treatment and advice as in group (A) in addition to low level laser therapy 3 session / week for 6 weeks.

All participants will be given a full explanation of the protocol of the study and an informed consent form will be signed by each female before participating in the study .

ELIGIBILITY:
Inclusion Criteria:

* Adolescent females have to meet the following criteria in order to participate in this study:

  * Suffering from Monosymptomatic nocturnal enuresis.
  * Their ages will range from 10-18 years.
  * Resistance to medical treatment (desmopressin acetate)

Exclusion Criteria:

* Adolescent Females with the following criteria will be excluded from this study:

  * Psychological or neurological disorders or other organic disorders.
  * Any chronic diseases.
  * Spinal cord abnormalities associated neurogenic bladder.
  * Evidence of urinary tract infection.
  * Ectopic ureter In addition, chronic constipation or encopresis.

Ages: 10 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2023-09-08 (Estimated); Study Completion 2023-09-08 (Estimated)

PRIMARY OUTCOMES:
bladder capacity | up to 6 weeks
  Sonography for bladder capacity. It will be used to determine bladder capacity for all participants before the beginning of the study for both groups, and at end of the study

SECONDARY OUTCOMES:
Maximum voided volume | up to 6 weeks
  will be measured in all participants. using a voiding diary over 4 days before starting therapy for each female in both group A and B and after the treatment program.
Frequency of bed wet | up to 6 weeks
  It will be used to determine the number of bed wet for each female in both group A and B before and after the treatment program.

CONTACTS AND LOCATIONS:
Overall Officials: Mai Mo Shehata, lecturer, Principal Investigator — faculty of physical therapy
Locations (1):
- Faculty of physical therapy, Giza, Egypt